CLINICAL TRIAL: NCT07026916
Title: A Single-Arm, Multicenter, Open-Label, Phase II Clinical Study to Evaluate the Efficacy, Safety/Tolerability, and Pharmacokinetic Characteristics of GFH375 Monotherapy in Patients With Previously Treated KRAS G12D Mutant Metastatic Pancreatic Cancer
Brief Title: A Phase II Study to Evaluate GFH375 in Patients With KRAS G12D Mutant Metastatic Pancreatic Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Adjustment of Product Development Strategy
Sponsor: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFH375X1201
Record Dates: First submitted 2025-06-03; First posted 2025-06-18 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GFH375 (Experimental)
  Interventions: Drug: GFH375

INTERVENTIONS:
Drug: GFH375 — GFH375 will be administered at the 600mg QD, orally, until disease progression or intolerable toxicity.

SUMMARY:
This is a multicenter, open-label, phase II study to explore the efficacy, safety/tolerability and pharmacokinetics (PK) of GFH375 in in Patients with Previously Treated KRAS G12D Mutant Metastatic Pancreatic Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form.
2. Male or female ≥ 18 years old and ≤75 years old.
3. With histologically or cytologically confirmed metastatic pancreatic cancer harboring KRAS G12D mutation
4. Be able to provide tumor tissue samples that meet the requirements
5. Have at least one measurable lesion according to RECIST1.1
6. ECOG performance status of 0-1.
7. With a life expectancy of ≥12 weeks.
8. Adequate laboratory parameters during the screening period.

Exclusion Criteria:

1. Active brain metastases.
2. Prior treatment with a KRAS G12D inhibitor or a pan-RAS/KRAS inhibitor.
3. With poorly controlled or severe cardiovascular disease.
4. Subjects with active hepatitis B or active hepatitis C.
5. Known allergy to the study drug or its components.
6. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 24 months
  ORR assessed by Blinded Independent Central Review

SECONDARY OUTCOMES:
ORR | 24 months
  ORR assessed by investigators
DCR | 24 months
  Disease control rate (DCR)
DoR | 24 months
  Duration of Response (DoR)
TTR | 24 months
  Time to Response(TTR)
PFS | 24 months
  Progression Free Survival (PFS)
The incidence and severity of AEs and SAEs | 24 months
  The incidence and severity of AEs and SAEs
Plasma concentrations of GFH375 | 6 months
  Plasma concentrations of GFH375

IPD SHARING:
Plan to Share IPD: No